CLINICAL TRIAL: NCT00509041
Title: A Phase II Study of Dasatinib (NSC #732517) in Patients With Previously Treated Malignant Mesothelioma
Brief Title: Dasatinib in Treating Patients With Previously Treated Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30601; U10CA031946 (NIH); CALGB-30601; CDR0000558362 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Results first posted 2013-01-17 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Malignant Mesothelioma
Keywords: advanced malignant mesothelioma; epithelial mesothelioma; recurrent malignant mesothelioma; sarcomatous mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib (Experimental): Use of dasatinib in treatment of pts with previously treated malignant mesothelioma
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — 50 mg PO bid

SUMMARY:
RATIONALE: Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well dasatinib works in treating patients with previously treated malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the rate of progression-free survival (PFS) at 24 weeks (or 5.5 months) in patients with malignant mesothelioma treated with dasatinib.

Secondary

* To determine the response rate (partial response [PR] and complete response [CR]) in patients with malignant mesothelioma treated with dasatinib.
* To determine the response duration in patients with malignant mesothelioma treated with dasatinib.
* To describe the overall survival (OS) of patients with malignant mesothelioma treated with dasatinib.
* To describe the toxicity profile of dasatinib in patients with malignant mesothelioma.
* To determine whether the amount of expression of EphA2 and PDGFRβ, as measured by immunohistochemistry from tumor specimens, correlates with PFS in patients with malignant mesothelioma.
* To determine whether plasma levels of VEGF and PDGFRβ, serum levels of CSF-1, and soluble mesothelin-related protein correlate with PFS in patients with malignant mesothelioma.
* To determine whether inhibition of Src phosphorylation in PBMC correlates with PFS.
* To assess inhibition of phosphorylation of Src, EphA2, and PDGFRβ in tumor tissue by dasatinib.

OUTLINE: Patients receive oral dasatinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood sample collection periodically for correlative studies. Tumor tissue samples are analyzed for EphA2 and PDGFRβ expression by immunohistochemistry. Tumor tissue samples may also be analyzed for phosphorylation of Src, EphA2, and PDGFRβ by western blot. Blood samples are analyzed for concentration of VEGF and PDGF by quantitative sandwich enzyme immunoassay technique; mesothelin-related protein level by Mesomark® assay; CSF-1 level by ELISA assay; and phosphorylation of Src by phospho-Src (pTyr418) human ELISA.

After completion of study treatment, patients are followed at least every 2 months for 1 year, then every 4 months for 1 year, then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant mesothelioma of any of the following subtypes:

  * Epithelial
  * Sarcomatoid
  * Mixed
* Any site of origin of malignant mesothelioma allowed including, but not limited to, any of the following:

  * Pleura
  * Peritoneum
  * Pericardium
  * Tunica vaginalis
* Pathology blocks or slides from a core surgical biopsy must be available
* Not amenable to curative surgery
* Measurable disease, defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques (CT scan , MRI, or x-ray) or as ≥ 10 mm with spiral CT scan

  * Patients with pleural rind only disease must have at least one level with one rind measurement ≥ 1.5 cm
  * Lesions that are considered nonmeasurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Prior treatment with one and only one systemic chemotherapy regimen, which must have included pemetrexed disodium required

  * Treatment may have been with pemetrexed disodium alone or in combination with any other agent
* No symptomatic pleural effusions, unless the patient undergoes a therapeutic thoracentesis

  * Patients with pleural effusions who have had a pleurodesis are eligible
* No known brain metastases
* May be registered on CALGB-150707 companion study

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Granulocytes ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Total bilirubin ≤ 2 x upper limit of normal (ULN)
* AST (SGOT) ≤ 2.5 x ULN
* Creatinine clearance ≥ 60 mL/min
* INR < 1.5
* PTT < 40 seconds
* QTc < 450 msec
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No significant cardiac disease, including any of the following:

  * New York Heart Association (NYHA) class III-IV congestive heart failure (CHF)
  * Unstable angina
  * Myocardial infarction or ventricular tachyarrhythmia within 6 months of study entry
  * Ejection fraction less than institutional normal (in patients with a history of CHF or currently with NYHA class I or II CHF)
  * Prolonged QTc > 450 msec (Fridericia correction)
  * Major conduction abnormality, unless a cardiac pacemaker is present
  * Hypokalemia or hypomagnesemia that cannot be corrected
* No history of significant bleeding disorder unrelated to cancer, including any of the following:

  * Congenital bleeding disorder (e.g., von Willebrand disease)
  * Acquired bleeding disorder within the past year (e.g., acquired anti-factor VIII antibodies)
  * Ongoing or recent (≤ 3 months) significant GI bleeding or hemoptysis
* No requirement for supplemental oxygen (i.e., pulse oximetry < 89% at rest)

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior pemetrexed disodium-containing chemotherapy
* At least 4 weeks since prior major surgery
* At least 4 weeks since prior radiation therapy

  * Measurable disease must be outside the radiation port
* Prior intracavitary cytotoxic or sclerosing therapy (including bleomycin) allowed

  * Intrapleural cytotoxic chemotherapy will not be considered systemic chemotherapy
* At least 7 days since prior and no concurrent antithrombotic or anti-platelet agents, including any of the following:

  * Aspirin or aspirin-containing combinations
  * Clopidogrel
  * Dipyridamole
  * Tirofiban
  * Epoprostenol
  * Eptifibatide
  * Cilostazol
  * Abciximab
  * Ticlopidine
  * Warfarin

    * Low-dose warfarin for prophylaxis to prevent catheter thrombosis allowed
  * Heparin or low molecular weight heparin

    * Heparin for IV line flush allowed
* At least 7 days since prior and no concurrent use of the following drugs:

  * Itraconazole
  * Ketoconazole (at doses > 200 mg/day)
  * Miconazole
  * Voriconazole
  * Telithromycin
  * Primidone
  * Rifabutin
  * Rifampin
  * St. John's wort
  * Carbamazepine
  * Oxcarbazepine
  * Rifapentine
  * Phenobarbital
  * Phenytoin
  * Quinidine
  * Procainamide
  * Disopyramide
  * Amiodarone
  * Sotalol
  * Ibutilide
  * Dofetilide
  * Erythromycin
  * Clarithromycin
  * Chlorpromazine
  * Haloperidol
  * Mesoridazine
  * Thioridazine
  * Pimozide
  * Bepridil
  * Droperidol
  * Halofantrine
  * Levomethadyl
  * Sparfloxacin
* No concurrent H2 blockers or proton pump inhibitors
* No bisphosphonate therapy during the first 8 weeks of study treatment
* No concurrent hormones or other chemotherapeutic agents except for steroids administered for dasatinib-related pleural effusion or hormones administered for non-disease-related conditions (e.g., insulin for diabetes)
* No concurrent palliative radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Dudek, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (37):
- United States (37):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Harry & Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - CCOP - Greenville, Greenville, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia

REFERENCES:
- [Result] Dudek A, Pang H, Kratzke RA, et al.: CALGB 30601: A phase II study of dasatinib (D) in patients (pts) with previously treated malignant mesothelioma (MM). [Abstract] J Clin Oncol 28 (Suppl 15) A-7037, 2010.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2007 to August 2009, 46 participants were recruited.
Pre-assignment Details: Three (3) participants withdrew from the study before treatment initiation; therefore 43 participants were eligible for evaluation
Groups:
- Dasatinib: Use of dasatinib (50 mg orally twice a day) in treatment of pts with previously treated malignant mesothelioma
Period: Overall Study
Arm/Group | Dasatinib
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 68 [35 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 43
ECOG Performance Score [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  participants
    0 - Fully Active | 19
    1 - Ambulatory, restricted strenuous activity | 24
Site of origin [Number; unit: participants]
  Pleura | 36
  Peritoneum | 6
  Other | 1
Histology [Number; unit: participants]
  Epithelial | 33
  Biphasic | 5
  Sarcomatoid | 2
  Not reported | 3
Prior chemotherapy [Number; unit: participants]
  Yes | 43
  No | 0
Prior radiation [Number; unit: participants]
  Yes | 6
  No | 37
Prior surgery [Number; unit: participants]
  Yes | 23
  No | 20

OUTCOME MEASURES:

1. Primary Outcome: 24 Week Progression Free Survival
Description: Percentage of participants who were alive and progression free at 24 weeks. The 24 week progression free survival, with 95% confidence interval, was estimated using the Kaplan Meier method.
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 43
percentage of participants | 23 [13.5 to 40]

2. Secondary Outcome: Number of Participants With Overall Tumor Response
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  * Complete Response (CR): disappearance of all target lesions;
  * Partial Response (PR) 30% decrease in sum of longest diameter of target lesions;
  * Progressive Disease (PD): 20% increase in sum of longest diameter of target lesions;
  * Stable Disease (SD): small changes that do not meet above criteria.
  Overall tumor response is the total number of CR and PRs.
Time Frame: Duration of study until progression (up to 3 years)
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 43
participants
  Complete Response | 0
  Partial Response | 2

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from registration to death of any cause. Surviving patients were censored at the date of last follow-up. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Time from registration to death (up to 3 years)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dasatinib
Number analyzed (Participants) | 43
weeks | 26.1 [18.6 to 36.7]

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) was defined as the time from registration to progression or death of any cause. Progression free and alive patients were censored at the date of last follow-up. The median PFS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Time from registration to progression or death (up to 3 years)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dasatinib
Number analyzed (Participants) | 43
weeks | 9.1 [7.4 to 16.9]

ADVERSE EVENTS:
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 15/43
Other Adverse Events (participants affected / at risk) | 35/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=43)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (11)
Pericardial effusion (Cardiac disorders) | 2 (2)
Watering eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8)
Peritoneal pain (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 10 (13)
Fever (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 3 (3)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (4)
Weight loss (Investigations) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (8)
Serum calcium decreased (Metabolism and nutrition disorders) | 6 (7)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 2 (2)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=43)
Hemoglobin decreased (Blood and lymphatic system disorders) | 24 (64)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 14 (19)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (19)
Stomach pain (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 6 (9)
Chest pain (General disorders) | 3 (5)
Chills (General disorders) | 3 (3)
Disease progression (General disorders) | 2 (2)
Edema limbs (General disorders) | 2 (7)
Fatigue (General disorders) | 24 (57)
Fever (General disorders) | 4 (5)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Visceral edema (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (2)
Upper aerodigestive tract infection (Infections and infestations) | 1 (3)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (5)
Alkaline phosphatase increased (Investigations) | 2 (6)
Aspartate aminotransferase increased (Investigations) | 3 (6)
Creatinine increased (Investigations) | 1 (1)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (9)
Platelet count decreased (Investigations) | 3 (3)
Weight loss (Investigations) | 7 (18)
Anorexia (Metabolism and nutrition disorders) | 11 (13)
Blood glucose increased (Metabolism and nutrition disorders) | 6 (10)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 5 (6)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (4)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 4 (4)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 10 (10)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (7)
Dysgeusia (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 8 (10)
Memory impairment (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Urogenital disorder (Renal and urinary disorders) | 1 (6)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (40)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (18)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (7)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes